CLINICAL TRIAL: NCT03635281
Title: Effect of Recruitment Maneuvers Plus Optimal PEEP Versus Optimal PEEP Alone on Ventilation Perfusion Mismatch and Respiratory Mechanics in One Lung Ventilation. A Randomized Trial
Brief Title: Effect of Recruitment Maneuvers Plus Optimal PEEP Versus Optimal PEEP Alone in One Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Professor, PhD, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OLVRM
Record Dates: First submitted 2018-07-31; First posted 2018-08-17 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEP group (Experimental): In this group the a PEEP level will be added after 20 minutes from OLV. PEEP values will be chosen according to the best static compliance with an incremental trial (i.e. starting from ZEEP, the PEEP values will be increased in step of 2 cmH2O each until the best compliance is reached)
  Interventions: Procedure: incremental PEEP
- RM+PEEP group (Experimental): Recruitment maneuvers will be performed as follow Recruitment maneuvers
  1. set FIO2 at 1.0
  2. Ppeak limit at 45 cmH2O
  3. Respiratory rate set at 6
  4. I:E set at 1:1
  5. Raise the VT at step of 2 ml/kg PBW until the Pplat is between 30-40 cmH2O
  6. If the maximum VT is set without rasing the Pplat, raise PEEP
  7. Allow three respiratory cycles with Pplat between 30 and 40 cmH2O
  8. End of RM
  The recruitment manouvers will be performed after 20 minutes of OLV. At the end of the RM, the VT will be set back to 5 ml/kg while the PEEP will be chosen according to the best static compliance with a decremental trial (from 16 cmH2O, lowering PEEP with steps of 2 cmH2O each until the best compliance is reached).
  Interventions: Procedure: Recruitment manoeuvers

INTERVENTIONS:
Procedure: Recruitment manoeuvers — Recruitment manoeuvers will be performed as follow Recruitment manoeuvers
  1. set FIO2 at 1.0
  2. Ppeak limit at 45 cmH2O
  3. Respiratory rate set at 6
  4. I:E set at 1:1
  5. Raise the VT at step of 2 ml/kg PBW until the Pplat is between 30-40 cmH2O
  6. If the maximum VT is set without rasing the Pplat, raise PEEP
  7. Allow three respiratory cycles with Pplat between 30 and 40 cmH2O
  8. End of RM
  The recruitment manouvers will be performed after 20 minutes of OLV. At the end of the RM, the VT will be set back to 5 ml/kg while the PEEP will be chosen according to the best static compliance with a decremental trial (from 16 cmH2O, lowering PEEP with steps of 2 cmH2O each until the best compliance is reached).
  Arms: RM+PEEP group
Procedure: incremental PEEP — In this group the a PEEP level will be added after 20 minutes from OLV. PEEP values will be chosen according to the best static compliance with an incremental trial (i.e. starting from ZEEP, the PEEP values will be increased in step of 2 cmH2O each until the best compliance is reached
  Arms: PEEP group

SUMMARY:
The intraoperative driving pressure (∆P) has been recently identified as the greater independent predictor of postoperative pulmonary complications after one lung ventilation (OLV). The application of a positive end-expiratory pressure (PEEP) level of 5 or 10 cmH2O has been shown to reduce the ∆P and the V/Q mismatch (Spadaro 2017); however, the "optimal" PEEP level able to minimize the ∆P may change significantly across patients. The aim of this study is to describe the optimal PEEP levels in patients undergoing thoracic surgery

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing VATS with OLV ≥2 hours

Exclusion Criteria:

* ASA (American Society of Anesthesiologists Physical Status Classiﬁcation) score ≥ 4
* severe chronic respiratory failure (chronic obstructive pulmonary disease patients with GOLD stage 3 or 4
* preoperative hemoglobin less than 10 g ml-1
* hemodynamic instability (defined as a decrease in systolic arterial pressure of more than 20% from baseline),

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
pulmonary shunt, expressed as percentage, measured by ALPE system | 20 minutes after intervention

SECONDARY OUTCOMES:
intraoperative driving pressure, measured as plateau pressure - PEEP | 20 minutes after intervention

OTHER OUTCOMES:
intraoperative oxygenation, measured as PaO2/FIO2 ratio | 20 minutes after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Spadaro S, Grasso S, Karbing DS, Fogagnolo A, Contoli M, Bollini G, Ragazzi R, Cinnella G, Verri M, Cavallesco NG, Rees SE, Volta CA. Physiologic Evaluation of Ventilation Perfusion Mismatch and Respiratory Mechanics at Different Positive End-expiratory Pressure in Patients Undergoing Protective One-lung Ventilation. Anesthesiology. 2018 Mar;128(3):531-538. doi: 10.1097/ALN.0000000000002011. PMID 29215365
- [Derived] Spadaro S, Grasso S, Karbing DS, Santoro G, Cavallesco G, Maniscalco P, Murgolo F, Di Mussi R, Ragazzi R, Rees SE, Volta CA, Fogagnolo A. Physiological effects of two driving pressure-based methods to set positive end-expiratory pressure during one lung ventilation. J Clin Monit Comput. 2021 Oct;35(5):1149-1157. doi: 10.1007/s10877-020-00582-z. Epub 2020 Aug 20. PMID 32816177